CLINICAL TRIAL: NCT01828125
Title: A Double-blinded, Randomized, Two-way, Cross-over Study to Assess the Efficacy of Small Subcutaneous Glucagon Dose Against the Conventional 1 mg Dose to Treat Hypoglycemia in Adults With Type 1 Diabetes
Brief Title: Efficacy of Small Subcutaneous Glucagon Dose to Treat Hypoglycemia in Adults With Type 1 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mini-doses glucagon
Record Dates: First submitted 2013-04-02; First posted 2013-04-10 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Glucagon; Hypoglycaemic hyperinsulinemic clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperinsulinemic hypoglycaemic clamp 1mg glucagon (Active Comparator): A 1.0mg glucagon dose will be given during the hyperinsulinemic hypoglycaemic clamp
  Interventions: Procedure: Hypoglycaemic hyperinsulinemic clamp; Drug: Glucagon
- Hyperinsulinemic hypoglycaemic clamp 0.1 or 0.2mg glucagon (Active Comparator): A dose of 0.1mg or 0.2mg will be given during the hyperinsulinemic hypoglycaemic clamp.
  Interventions: Procedure: Hypoglycaemic hyperinsulinemic clamp; Drug: Glucagon

INTERVENTIONS:
Procedure: Hypoglycaemic hyperinsulinemic clamp — A first catheter will be inserted for infusion of D-[6,6-2H2] glucose and insulin. A second catheter will be inserted for infusion of dextrose. Dextrose infusion will be enriched with D-[6,6-2H2] glucose. A third catheter will be inserted for sampling. D-[6,6-2H2] glucose will be administered as a priming dose followed by a constant infusion throughout the experiment. Insulin will be administered as a primed continuous infusion. The first two hours will serve as an equilibration period for the tracer while glucose infusion will be adjusted to achieve a plasma glucose concentration of 5 mmol/L. The third hour is considered the baseline period. Following this, dextrose infusion rate will be decreased over a period of 1 hour to attain hypoglycaemia with a target blood glucose level at 2.8 mmol/L. At the end of the fourth hour, a subcutaneous glucagon dose will be given and plasma samples will be drawn for the determination of labelled and unlabelled glucose, plasma insulin and glucagon.
Drug: Glucagon

SUMMARY:
In the unfortunate case of severe hypoglycaemia, glucagon is the first-line treatment because of its potent and rapid action starting as fast as 5 minutes after subcutaneous or intramuscular injection. Large dose of glucagon such as 1 mg subcutaneous is usually associated with undesirable side-effects such as nausea, vomiting, bloating and headache.

The overall objective of this research proposal is to assess the efficacy of lower subcutaneous doses of glucagon (0.1 mg or 0.2 mg) to correct hypoglycaemia compared to the standard dose (1.0 mg) in adults with type 1 diabetes mellitus (T1D).

It is postulated that much lower dosages of glucagon (0.1 or 0.2 mg) injected subcutaneously will be just as effective as the current recommended dose of 1.0 mg to correct hypoglycaemia without the undesirable gastro-intestinal side effects.

DETAILED DESCRIPTION:
In the unfortunate case of severe hypoglycaemia, glucagon is the first-line treatment because of its potent and rapid action starting as fast as 5 minutes after subcutaneous or intramuscular injection. Current instructions for the treatment of severe hypoglycaemia call for the immediate injection of 1 mg of glucagon subcutaneously or intramuscularly. Large dose of glucagon such as 1 mg subcutaneous is usually associated with undesirable side-effects such as nausea, vomiting, bloating and headache. Moreover, glucagon emergency kits are relatively expensive (around $100 per kit), thus increasing the financial burden of diabetes on patients and the health care system.

The primary objective of this research project is to the study the pharmacological effects of different doses of glucagon injected subcutaneously to correct hypoglycaemia during controlled conditions mimicking a hypoglycaemic event in adults with type 1 diabetes. More specifically, we will be looking at the effects of subcutaneous glucagon injected at 0.1 or 0.2 mg and 1.0 mg to normalized plasma glucose during a hypoglycaemic hyperinsulinemic clamp in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of old
* Clinical diagnosis of type 1 diabetes for at least two years.

Exclusion Criteria:

* Clinically significant nephropathy (MDRD < 60 mL/min/1.73 m2).
* Pregnancy
* Severe hypoglycemic episode within two weeks of screening
* Current use of glucocorticoid medication (except low stable dose)
* Pheochromocytoma or primary adrenal insufficiency (e.g. Addison's disease)
* Medical condition likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Incremental area under the curve of plasma glucose concentrations | 30 minutes
  30-min incremental area under the curve of plasma glucose concentrations starting at the time glucagon is injected subcutaneously

SECONDARY OUTCOMES:
Time to reach glucose levels ≥ 4 mmol/L | Up to 2.5 hours
Time to reach glucose levels ≥ 5 mmol/L | Up to 2.5 hours
Time-to-peak plasma glucagon concentration | Up to 2.5 hours
  Time-to-peak plasma glucagon concentration after glucagon injection
Time for 25% of glucagon appearance | Up to 2.5 hours
  Time for 25% of glucagon appearance after glucagon injection
Time for 50% of glucagon appearance | Up to 2.5 hours
  Time for 50% of glucagon appearance after glucagon injection
Time for 75% of glucagon appearance | Up to 2.5 hours
  Time for 75% of glucagon appearance after glucagon injection

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada